CLINICAL TRIAL: NCT01240070
Title: Multicenter, Randomized Trial Designed to Evaluate the Applicability of the Guidelines of the Italian Society of Diabetology for the Prevention of Cardiovascular Diseases in Type 2 Diabetes
Brief Title: Multifactorial Intervention in Type 2 Diabetes - Italy
Acronym: MINDIT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Parma (Other)
Collaborators: Italian Society of Diabetology (Other); AstraZeneca (Industry); Daiichi Sankyo (Industry)
Responsible Party: FoRiSID, Research Foundation of the Italian Society of Diabetology, Italian Society of Diabetology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MINDIT2000
Record Dates: First submitted 2010-11-12; First posted 2010-11-15 (Estimated); Last update posted 2011-08-12 (Estimated); Status verified 2010-10

CONDITIONS: Type 2 Diabetes
Keywords: diabetes,; cardiovascular; risk factor; cardiovascular event; intervention
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Critical Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Care (Active Comparator): Clinical practice in type 2 diabetes treatment
  Interventions: Other: Intensive care
- Intensive Care (Active Comparator): Intensive multi-factorial treat-to-target intervention, according to international guidelines, that includes both lifestyle intervention and a step-wise strategy for pharmacological treatment with a treat-to-target approach.
  Interventions: Other: Intensive care

INTERVENTIONS:
Other: Intensive care — Intensive multi-factorial treat-to-target intervention program designed according to international guidelines

SUMMARY:
Despite several clinical trials have clearly demonstrated that the correction of a single cardiovascular risk factor in patients with type 2 diabetes decreases the incidence of myocardial infarction and other cardiovascular disease (CVD) events, only the Steno study has been evaluating the effect of a multifactorial intervention strategy on macrovascular complications of diabetes. For this reason, the disease management approach currently endorsed by international guidelines (i.e correction of all major CVD risk factors to target levels usually lower than lower risk populations) has not been extensively investigated in terms of prevalence of application in current clinical practice and in terms of real efficacy.

The Multifactorial INtervention in type 2 Diabetes - ITaly (MIND.IT) is a multicentric two-phase study involving 9 Diabetes Care Units throughout Italy with the overall aims of: (1) investigating the degree of application of the international guidelines for CVD prevention in type 2 diabetic patients and (2) verifying whether the application of an intensive multi-factorial intervention inspired by these guidelines is feasible and effective in decreasing the incidence of new CVD events.

DETAILED DESCRIPTION:
The study is multi-centric, randomized, open label, active treatment controlled, two parallel-group, pragmatical intervention trial with 5 years of follow-up, to assess superiority of an intensive treat-to-target strategy (including lifestyle and pharmacological interventions) for correction of major cardiovascular risk factors compared to usual care in decreasing incidence of first cardiovascular events in non complicated type 2 diabetic patients at high risk, as defined by presence of 2 or more cardiovascular risk factors. All high-risk patients identified during phase 1 who accepted to participated were allocated to usual or intensive treatment based on the recruiting center. Centers were randomly assigned to treatment arm before phase 2 beginning. Investigators from Intensive Care centers received centralized training to ensure the application of the intensive care program on their patients.

HbA1c values and lipid profile are assessed in peripheral laboratories (one per each study site) with an external, centralized, quality control program and the adjustment for systematic differences among study labs.

Participating investigators are left free to decide upon patient's treatments. In intensive-care centers, investigators are provided with a multi-factorial step-wise protocol to support the application of a treat-to-target approach. Intensive care strategy includes intervention on lifestyle.

Dietary intervention goals: BMI<25 or 5% reduction of body weight; dietary assumption of saturated fat <10% of total caloric intake; fibers= 15-20 g/1000 Kcal. Methods defined to reach the dietary goal: A) Patients with BMI 25-30 kg/m2: reduction of caloric intake = 300-500 Cal/d; B) Patients with BMI >30: reduction of caloric intake 500-800 Cal/d.

Physical activity intervention goal: 200-300 calories per day. Example: brisk walking for 30 min every day or biking (18-25Km/h 45-60 min). Alternatives: swimming 1h , dancing 1h, gym exercise 1h;-avoiding isometric exercise and exercise with intensity >50-60 % of maximal oxygen consumption. Frequency: everyday or at least 3 times a week; Pharmacological intervention: Blood glucose control, multi-step intervention. In obese patients: 1) Metformin (M, 500-2500mg); 2) M+Sulphonylureas (S) or S-like drugs, increasing progressively the dose; 3) M+S+Acarbose; 4) M+S+insulin bed-time; 5) insulin basal-bolus. In normal weight patients: 1) S; 2) S+acarbose; 3) S+ bed-time insulin; 4) insulin basal bolus; Blood pressure control --> 1) Ace-inhibitors or AT-II receptor antagonists; 2) add long acting calcium-channel blockers or beta-blockers or low dose diuretics; 3) add a third drug; lipid control: 1) diet + physical activity; 2) if LDL > 130 mg/dL statins (with a stepwise increase of dose if necessary); if triglycerides > 200 mg/dL fibrates; anti-platelet treatment: aspirin 100 mg/d in all patients (alternative drugs for aspirin-intolerants).

The scheduled visits were defined as follows:

* Intensive-care group: mandatory visit every three months with annual visit for MIND.IT data collection.
* Usual-care group: at least one MIND.IT visit every year + the usual organization of the center.

ELIGIBILITY:
Inclusion Criteria:

* Both genders
* age 50-70 years
* Type two diabetes with at least two-year history of disease and without insulin treatment in the first two years after diagnosis
* Negative medical history for documented previous cardiovascular events or macrovascular complications
* Written consent to participate
* Presence of at least 2 of the following risk factors:

  * LDL cholesterol > 130 mg/dL (regardless of treatment)
  * Triglycerides > 200 mg/dL
  * HDL cholesterol < 35 (males) or 45 (females) mg/dL
  * Blood pressure > 140/90 mmHg
  * Cigarette smoking

Exclusion Criteria:

* Age below 50 or above 70 years
* Type 1 diabetes, diagnosis before 40 years of age, known presence of auto-antibodies or insulin requirement in the first 2 years of disease.
* Chronic kidney failure (plasma creatinine > 2 mg/dL)
* Significant liver damage (AST and/or ALT > 2 times the upper limits of normality)
* History of previous cardiovascular events
* Active neoplasms or any concomitant disease limiting life expectancy

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1461 (Actual)
Dates: Start 2002-01; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular events | 5 years of follow up
  To verify if an intensive care intervention compared to usual care is able to significantly decrease the incidence of first cardiovascular event. Composite primary end-point = mortality for cardiovascular causes, proven acute myocardial infarction (STEMI or NSTEMI), acute coronary syndrome requiring hospitalization, proven ischemic stroke, coronary or carotid revascularization procedure

SECONDARY OUTCOMES:
cardiovascular risk factors changes | 2 years and 5 years of follow up
  To assess whether the intensive treatment is able to significantly improve cardiovascular risk factors with increased multiple-target achievement. A pre-planned interim analysis after two years of follow-up was foreseen by the study protocol.
  To verify that the intesive protocol implemented on the basis of national and international guidelines is actually feasible in a real world clinical setting.

CONTACTS AND LOCATIONS:
Overall Officials: Ivana Zavaroni, MD, Study Chair — University of Parma; Angela A Rivellese, MD, Study Director — Federico II University of Naples; Olga Vaccaro, MD, Study Director — Federico II University of Naples; Roberto Miccoli, MD, Study Director — University of Pisa; Mariella Trovati, MD, Study Director — University of Turin, Italy; Franco Cavalot, MD, Study Director — University of Turin, Italy; Massimo Boemi, MD, Study Director — INRCA of Ancona; PierPaolo DeFeo, MD, Study Director — University Of Perugia
Locations (9):
- Italy (9):
  - Francesco Giorgino, Bari
  - Maria Dolci, Carrara
  - Lamberto De Giorgio, La Spezia
  - Giuseppe Derosa, Pavia
  - PierPaolo DeFeo, Perugia
  - Donatella Zavaroni, Piacenza
  - Roberto Miccoli, Pisa
  - Giovanni Ghirlanda, Roma
  - Mariela Trovati, Torino

REFERENCES:
- [Background] Rivellese AA, Boemi M, Cavalot F, Costagliola L, De Feo P, Miccoli R, Patti L, Trovati M, Vaccaro O, Zavaroni I; Mind.it Study Group. Dietary habits in type II diabetes mellitus: how is adherence to dietary recommendations? Eur J Clin Nutr. 2008 May;62(5):660-4. doi: 10.1038/sj.ejcn.1602755. Epub 2007 Apr 11. PMID 17426738
- [Background] Vaccaro O, Boemi M, Cavalot F, De Feo P, Miccoli R, Patti L, Rivellese AA, Trovati M, Ardigo D, Zavaroni I; MIND-IT Study Group. The clinical reality of guidelines for primary prevention of cardiovascular disease in type 2 diabetes in Italy. Atherosclerosis. 2008 Jun;198(2):396-402. doi: 10.1016/j.atherosclerosis.2007.10.026. Epub 2008 Feb 21. PMID 18093594
- [Derived] Vaccaro O, Franzini L, Miccoli R, Cavalot F, Ardigo D, Boemi M, De Feo P, Reboldi G, Rivellese AA, Trovati M, Zavaroni I; MIND.IT Study Group. Feasibility and effectiveness in clinical practice of a multifactorial intervention for the reduction of cardiovascular risk in patients with type 2 diabetes: the 2-year interim analysis of the MIND.IT study: a cluster randomized trial. Diabetes Care. 2013 Sep;36(9):2566-72. doi: 10.2337/dc12-1781. Epub 2013 Jul 17. PMID 23863908
- [Derived] Ardigo D, Vaccaro O, Cavalot F, Rivellese AA, Franzini L, Miccoli R, Patti L, Boemi M, Trovati M, Zavaroni I; MIND.IT study group. Effectiveness of treat-to-target strategy for LDL-cholesterol control in type 2 diabetes: post-hoc analysis of data from the MIND.IT study. Eur J Prev Cardiol. 2014 Apr;21(4):456-63. doi: 10.1177/2047487312467746. Epub 2012 Nov 12. PMID 23147277